CLINICAL TRIAL: NCT05639322
Title: Psychotherapy for Ketamine's Enhanced Durability in Chronic Neuropathic Pain: A Randomized Controlled Pilot Trial
Acronym: PSYKED-NP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: P-003
Record Dates: First submitted 2022-11-28; First posted 2022-12-06 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-10

CONDITIONS: Neuropathic Pain
Keywords: Feasibility trial; Ketamine; Cognitive behavioural therapy
MeSH Terms: conditions — Neuralgia | interventions — Ketamine; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ketamine only (Active Comparator)
  Interventions: Drug: Ketamine Hydrochloride
- Psychotherapy only (Active Comparator)
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Ketamine + Psychotherapy (Experimental)
  Interventions: Other: Ketamine + Cognitive Behavioral Therapy

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Ketamine-HCL IV 1mg/kg (up to 100 mg) over 2 hours, on weeks 2, 7, and 12.
  Arms: Ketamine only
Behavioral: Cognitive Behavioral Therapy — Cognitive Behavioural Therapy/ Mindfulness Based Meditation therapy (CBT/MM) remotely for 16 hours between weeks 1 to 16 inclusive + in-person sessions on weeks 2, 7 and 12
  Arms: Psychotherapy only
Other: Ketamine + Cognitive Behavioral Therapy — Ketamine-HCL + CBT/MM according to the same directions specified in Arm 1 and Arm 2.
  Arms: Ketamine + Psychotherapy

SUMMARY:
The purpose of the study is to investigate new therapies to alleviate pain on neuropathic chronic pain. At this time, the main purpose is to complete a feasibility or pilot study with 60 participants suffering from neuropathic chronic pain. Participants will be randomized to (1) Ketamine (Hydrochloride) HCL; (2) psychotherapy (using Cognitive Behavioral Therapy); or (3) a combination of Ketamine HL and psychotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age
2. Diagnosis of chronic neuropathic pain as determined by a pain specialist with moderate-to-severe neuropathic pain as per ID pain questionnaire, with mean pain scores > 3 on a numeric rating scale (NRS), in the 7 days preceding inclusion
3. For participants of childbearing potential, use highly effective or double-barrier methods of contraception. Abstinence is acceptable if it is the preferred and usual lifestyle of the participant
4. Capacity to provide informed consent

Exclusion Criteria:

1. Patients less than 18 years of age
2. Current or lifetime history of schizophrenia, psychotic disorder, bipolar disorder, or borderline personality disorder
3. Known history of hypersensitivity or allergy to Ketamine-HCL
4. Current history of dissociative disorders
5. Current concomitant use of theophylline or aminophylline
6. Current elevated intracranial pressure
7. Pregnancy or ongoing breastfeeding in female participants
8. Concomitant active substance use in the 6 months preceding enrolment (amphetamines, alcohol, and ketamine)
9. Contraindication to receiving Ketamine-HCL (e.g. current or lifetime history of cerebrovascular accident; current significant hypertension [systolic blood pressure higher than 160 mmHg and/or diastolic blood pressure higher than 100 mmHg]; current severe cardiac decompensation [e.g. presence of dyspnea, peripheral edema, elevated jugular venous pressure, hepatomegaly, pulmonary rales, pleural effusions])

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2025-07-24 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 2 years
  Recruitment rate and withdrawal rate (Acceptability and feasibility study)
Adherence rate | 2 years
  Feasibility
Frequency of adverse events | 2 years
  Safety and tolerability

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System Pain Interference (PROMIS) Pain Intensity, 1 a. | 20 weeks
  PROMIS-PI - 1 a. pain intensity scale- 0 to 10 (The higher the number the higher the pain intensity)
Patient-Reported Outcomes Measurement Information System Pain Interference, PROMIS 6 a. Pain Interference, | 20 weeks
  PROMIS-PI -Short form 6 a. - pain interference scale- 6 items, 5 likert scale The higher the score the higher the interference from pain)

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No individual participant data has been planned to be shared with other researchers at this point, since this is a feasibility study with only 60 participants

REFERENCES:
- [Derived] Goel A, Kapoor B, Chan H, Ladha K, Katz J, Clarke H, Pazmino-Canizares J, Thomas Z, Philip K, Mattina G, Ritvo P. Psychotherapy for Ketamine's Enhanced Durability in Chronic Neuropathic Pain: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2024 Apr 17;13:e54406. doi: 10.2196/54406. PMID 38630524